CLINICAL TRIAL: NCT05194631
Title: Evaluation of the Regeneration Capacity of Satellite Cells From the Quadriceps Compared to That of the Diaphragm
Acronym: ECARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL21_0384
Record Dates: First submitted 2021-12-09; First posted 2022-01-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-08

CONDITIONS: Diaphragm Injury; Mechanical Ventilation Complication
Keywords: Satellite cells; mechanical and oxidative stress; regenerative function

STUDY DESIGN:
Intervention Model Description: This is a prospective cross-sectional study involving category humans, which aims is to assess the pathophysiological mechanisms of a deficit in muscle fiber regeneration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regeneration Capacity of Satellite Cells (Experimental): In vitro Regeneration Capacity of Satellite Cells from the Quadriceps Compared to That of the Diaphragm isolated From one patient
  Interventions: Other: Quadriceps microbiopsy using a Tru-Cut biopsy needle

INTERVENTIONS:
Other: Quadriceps microbiopsy using a Tru-Cut biopsy needle — During surgery for a benign or malignant tumor of the liver a quadriceps microbiopsy will be performed. A 1 cm incision of the skin and fat planes will be made using a scalpel until contact with the quadriceps aponeurosis. The biopsy needle will be inserted superficially into the muscular part allowing, through a suction system, a micro biopsy of the quadriceps of approximately 25 mg.

SUMMARY:
Actually no treatment exists to prevent the loss of diaphragmatic function induced by mechanical ventilation during an intensive care unit stay. The consequence is a growing number of survivors with moderate to severe chronic respiratory disease so called Ventilation-Induced Diaphragmatic Dysfunction (VIDD). This study complements the BOTAN study (IRB Accreditation number: 198711, NCT02900300) on 24/11/2021 under number 2021_IRB-MTP_08-37), which aim was the constitution of a biological bank of diaphragmatic tissue in order to be able to propose an innovative tool for the in vitro screening of bioactive molecules of interest in human, to improve the regenerative capacity of this main and essential muscle for breathing. In this present study, in order to offer this evaluation tool in the screening of bioactive molecules of interest, without the need of the diaphragm biopsy, but simply of the quadriceps, the investigators propose, by adding a quadriceps muscular biopsy to patients already included in BOTAN study, to compare the regenerative capacity of quadriceps and diaphragmatic muscle in the same individual. Thus, this study is the first, which will propose a new minimally invasive tool for the evaluation and optimization of future pharmacological treatments targeted to limit the impact of VIDD.

Thus our main objective of thus study is to compare in the same patient the regenerative capacity of the muscular fiber of the quadriceps to that of the diaphragm in order to set up an in vitro model allowing to test in humans future pharmacological treatment devoted to limit the incidence of VIDD.

In this study will be recruited patients treated surgically for a benign or malignant tumor of the liver requiring surgical excision in contact with the diaphragm and who have agreed to participate in the BOTAN study. The resection to be complete (R0) must pass within the diaphragmatic muscle allowing us to obtain without any constraint for the patient, diaphragmatic tissue.

The provision of 10 samples will enable us to produce the cell cultures needed to achieve the study objectives. In order to take into account subjects who leave the study without meeting the primary endpoint, we plan to include up to 15 subjects.

During this surgery, for the purposes of the present study, the investigators will perform a quadriceps biopsy. Quadriceps biopsies are widely used in biomedical research and no deleterious effects have been described. The surgical team is fully qualified for this type of sampling and all experiments necessary to compare regenerative capacity of quadriceps and diaphragmatic muscular fiber use laboratory techniques perfectly mastered by our research team.

For each patients, this study will be performed over two visits. The first, during a consultation will allow the inclusion of the patient, as well as the collection of clinical data and a second during the scheduled surgical intervention where quadriceps biopsy will be realised. The expected duration of inclusions will be one year.

No immediate individual benefit is expected for the patient. This study aims to improve, in the future, therapies that reduce the incidence of diaphragmatic dysfunction induced by mechanical ventilation. In fact, diaphragmatic dysfunction induced by ventilation is observed in at least 50% of patients in intensive care; this dysfunction has been implicated in the significant lengthening of the hospital stay, the difficulties in weaning from mechanical ventilation and in the increased risk of co-morbidity and mortality. The validation of the first in vitro model in humans of this dysfunction, from quadriceps biopsy, will allow us to pre-select antioxidant molecules and the most effective concentrations to use for a future therapeutic trial aimed at limiting the deleterious effects of mechanical ventilation on the diaphragm in humans.

DETAILED DESCRIPTION:
This study focuses on mechanical ventilation used in intensive care unit to supplement ventilatory function in patients. Indeed, mechanical ventilation can "paradoxically" be at the origin of complications that can be life-threatening in patients. Indeed, mechanical ventilation buy unloading respiratory muscles, mays induce atrophy of these muscles and an alteration of their contractile properties induced by a disturbance of the redox status and tissue regeneration. This muscular pathology is called ventilation-induced diaphragmatic dysfunction (DDIV).

In animal models, antioxidant molecules showed a beneficial effect to limit this pathology, highlighting the importance of oxidative stress in the pathophysiology of DDIV. Among the different molecules tested, SS-31, which is a chelator of free radicals specific to the mitochondria, has shown its effectiveness in preventing VIDD in an animal model. However, physiopathological data in Human are still needed to propose this molecule in a therapeutic trial. Indeed, the maintenance of muscle mass and therefore tissue regeneration depends on the ability of muscle stem cells (MuSC) or satellite cells to activate and differentiate. Muscular homeostasis depends also on the capacity of these cells to activate quiescence genes in order to maintain a pool of quiescent cells which keep capacity for self-renewal. In the context of a pathological microenvironment favoring excessive activation of satellite cells, such as during mechanical ventilation, the investigators can postulate that this will lead to a loss of the pool of quiescent cells, thus inducing a loss of homeostasis of the muscle tissue responsible for long-term atrophy. Recent studies on mice, have shown a higher potential for these diaphragmatic quiescent cells to be activated and participating in the renewal of damaged muscle fibers in comparison to peripheral muscles. This specificity of early activation of diaphragmatic satellite cells could weaken them against a pathological microenvironment induced by mechanical ventilation, altering their regenerative capacity. But no data currently exists in humans.

The investigators therefore want, in this study, to assess the diaphragm specificity of the physiopathological mechanisms involved in VIDD, by a comparative study in the same subject of the biological function of satellite stem cells originating from the quadriceps muscle and the diaphragm. This study is complementary to the BOTAN project validated by the IRB of Montpellier (IRB Accreditation number: 198711), on 24/11/2021 under number 2021_IRB-MTP_08-37, allowing the collection of diaphragmatic satellite cells from the care. In fact, in subjects included in the BOTAN study, the investigators will perform, during the same surgical intervention, allowing access to a diaphragmatic biopsy, a biopsy of the quadriceps in order to evaluate in parallel the regenerative capacities of the stem cells of the quadriceps, compared to that of the diaphragm in the same patient.

Our hypothesis is that the mechanical and oxidative stress imposed by mechanical ventilation will lead to impaired activation of satellite cells, depletion of the pool of quiescent satellite cells. The consequence will be an inability of muscular tissue regeneration and ultimately atrophy associated diaphragm contractile dysfunction. Thus by comparing the biological function of satellite cells and their regenerative capacities coming from diaphragm and quadriceps of the same patient, the investigators will be able to answer the question of whether diaphragmatic stem cells are more active in their renewal compared to those of the quadriceps and therefore more likely susceptible to lose their pool of quiescent cells, at the basis of muscle atrophy and VIDD.

This work would allow us in the future to identify new therapeutic targets aimed at limiting the early activation of satellite cells at rest, harmful for the maintenance of a pool of quiescent satellite cells during mechanical ventilation, in order to limit the impact of the VIDD.

Moreover, the BOTAN study will allow us to propose a in vitro model of VIDD from cultures of human diaphragmatic stem cells, which will be subjected to mechanical stress similar to those encountered in ventilated patients. Thanks to the present study, which will allow us to assess the specificity of early activation of the quadriceps satellite cells compared to that of the diaphragm in the same individual, the investigators will also be able to validate a in vitro tool allowing the screening of bioactive molecules of interest to limit VIDD, without the need for a diaphragm biopsy but only a quadriceps biopsy, which is much more simple and less invasive. Thus, this study is the first study in humans to propose this type of comparative evaluation, which will make it possible to propose new minimally invasive tools in the evaluation and optimization of pharmacological treatments to limit the impact of VIDD.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 80 years old
* patient treated by the digestive surgery department of Montpellier University Hospital for a benign or malignant tumor of the liver requiring surgical excision in contact with the diaphragm who agreed to participate in the BOTAN study (Approval Number assigned by the IRB of Montpellier : 2021_IRB-MTP_08-37)
* patient clinically stable at the time of the study, ie not requiring any treatment

Exclusion Criteria:

* Patients undergoing treatment with antibiotics or corticosteroids, or recently within the last 4 months
* Pregnant or breastfeeding woman.
* Patients with a body mass index > 30
* Patients with any criteria that may in themselves impair respiratory muscle function such as chronic obstructive pulmonary disease, heart failure, systemic infection, neuromuscular pathology, psychiatric pathology or metabolic disorder.
* Patients with coagulopathy or thrombocytopenia.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the number and size of differentiating myoblasts obtained per satellite cells from the quadriceps with that of the diaphragm in the same patient | 3 months
  The quadriceps and diaphragm muscle biopsies will be placed in a culture dish treated with type 1 collagen in a thin layer of matrigel. 6 to 8 days later, the myoblasts are purified by MACS (Magnetic Activated Cell Sorting) based on the property of myoblasts to express the CD56 surface antigen. After culture on a collagen dish, proliferation and differentiation of the CD56 positive cells will be assessed by cell counting and immunofluorescence with antibodies directed against muscle markers.

SECONDARY OUTCOMES:
Elongation of muscle fibre length in a human model of ventilation-induced diaphragmatic dysfunction (VIDD) using myoblasts from the diaphragm and quadriceps | 3 months
  The myofibers obtained after satellite cells culture will be subjected to a protocol of elongation / shortening cycles mimicking the mechanical stresses induced in vivo during mechanical ventilation using a Flexcell®'s type device (FX-5000 ™ Tension System). The capacity of the systme to lengthen muscle fibre from the diaphragm and quadriceps will be assessed by fluorescence images acquired with Olympus microscope equipped with monochrome camera..
Evaluation of mechanical stresses of muscle fibres from the quadriceps and the diaphragm in a human model of ventilation-induced diaphragmatic dysfunction (VIDD) | 3 months
  The myofibers obtained after satellite cells culture will be subjected to a programme of stretching muscle fibres by 15% of their initial size at a frequency of 1 HZ for 24 hours using a Flexcell®'s type device (FX-5000 ™ Tension System).The induction of mechanical stresses will be assessed by chemiluminescence identification of a production of oxygen-reactive species and by evaluation of calcium homeostasis with Ca2+ Sparks Measurements using fluorescent calcium indicator (Fluo-3) and confocal microscopy. Results obtained will be compared between diaphragm and quadriceps.
Evaluation of the in vitro efficacy in humans of a mitochondria-specific anti-oxidant (SS-31) to prevent a deficit in muscle regeneration induced by oxidative stress | 3 months
  Assessment of oxygen-reactive species production by satellite cells cultured in medium containing SS-31 and subjected to a programme of stretching muscle fibres by 15% of their initial size at a frequency of 1 HZ for 24 hours using a Flexcell®'s type device (FX-5000 ™ Tension System) compared with a group of untreated cells in both diaphragm and quadriceps muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No